CLINICAL TRIAL: NCT00641316
Title: A Prospective Study of Bone Augmentation Techniques in Extraction Sockets and Implant Surface Textures
Brief Title: An Assessment of Bone Augmentation in Post-Extraction Sockets
Acronym: FMD-007
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: BioHorizons, Inc. (Industry)
Responsible Party: Principal Investigator, Nicolaas C. Geurs, DDS, MS, Department Chair, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F071006001
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Results first posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Unrestorable Dentition; Post-Extraction Sockets
Keywords: Freeze-dried bone allograft; Platelet-rich plasma; Platelet-derived growth factors; Laser-threaded dental implants; Resorbable blast textured dental implants
MeSH Terms: interventions — Transplantation, Homologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Teeth extraction followed by natural healing
  Interventions: Procedure: AtraumaticTeeth Extraction
- 2- FDBA/TCP (Experimental)
  Interventions: Procedure: Atraumatic Teeth Extraction/Grafted Extraction Sockets
- 3 FDBA/TCP+PRP (Experimental)
  Interventions: Procedure: Atraumatic Teeth Extraction/Grafted Extraction Sockets
- 4 FDBA/TCP + PDGF (Experimental)
  Interventions: Procedure: Atraumatic Teeth Extraction/Grafted Extraction Sockets

INTERVENTIONS:
Procedure: AtraumaticTeeth Extraction — Teeth extraction alone, allowed to heal for 2 months followed by implant therapy to the sites
  Other Names: Post-extraction socket healing
  Arms: 1
Procedure: Atraumatic Teeth Extraction/Grafted Extraction Sockets — Teeth extraction/post-extraction socket grafting with Freeze-Dried Bone Allograft (FDBA) mixed with Tri-Calcium Phosphate(TCP) allowed to heal for 2 months followed by dental implant therapy to the sites
  Other Names: Allograft
  Arms: 2- FDBA/TCP
Procedure: Atraumatic Teeth Extraction/Grafted Extraction Sockets — Teeth extraction/post-extraction socket grafting with FDBA/TCP enriched with Autologous Platelet-Rich Plasma (PRP) allowed to heal for 2 months followed by dental implant therapy to the sites
  Other Names: Platelet-rich plasma
  Arms: 3 FDBA/TCP+PRP
Procedure: Atraumatic Teeth Extraction/Grafted Extraction Sockets — Teeth extraction/post-extraction socket grafting with FDBA/TCP enriched with Platelet-Derived Growth Factors (PDGF) allowed to heal for 2 months followed by dental implant therapy to the sites
  Other Names: GEM-21
  Arms: 4 FDBA/TCP + PDGF

SUMMARY:
When a tooth is extracted the ridge of bone that held the tooth in place begins to heal and over time new bone grows to fill the empty space left by the missing tooth. Sometimes this process works very well and new bone grows to completely fill the socket, at other times new bone fails to fill in the space completely and patients are left with uneven bone-fill.

Grafted extraction sockets may fill with bone faster and more evenly than those without grafts, allowing the dentist to have greater control over the healing process and to repair the area with dental implants in a shorter period of time.

This study will help determine if grafting an extraction socket, with or without enriching the graft material, is an added benefit when compared to allowing the socket to heal naturally.

The study will also assess how well two different dental implant designs used to restore the area will function over time.

DETAILED DESCRIPTION:
Tooth extraction is often associated with resorption of the alveolar ridge height and width and with compromised soft tissue contours. A variety of methods have been proposed to overcome varied patterns of post-extraction healing.

An increasingly common practice combines skilled surgical technique with post-extraction site grafting utilizing both natural and synthetic bone-graft materials. These procedures are thought to retard resorption of the socket volume while lending some control over bone-fill - thereby preserving the integrity of the alveolar ridge for future reconstruction with dental implants.

Limited evidence-based data exist to support a variety of bone-graft materials including grafts enriched with autologous platelet-rich plasma(PRP)and grafts enriched with recombinant human platelet-derived growth factors(PDGF). Despite emerging clinical acceptance the most efficacious intervention remains undetermined.

In an effort to establish clinical evidence, this study will assess the efficacy of ridge preservation using three different bone grafting applications in post-extraction sockets compared to extraction alone.

The study will also asses longitudinal success of restoring the study sites with dental implants. Two innovative dental implant designs will be used in the study; an implant with a resorbable blast textured(RBT)surface and an implant with a laser thread-textured (LTT)surface.

ELIGIBILITY:
Inclusion Criteria:

* Needed extraction of Maxillary and/or Mandibular Incisors and/or Pre-molar teeth

Exclusion Criteria:

* Inability to provide informed consent in English
* Pregnant women

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Reddy, DMD, DMSc, Principal Investigator — University of Alabama at Birmingham; Nicolaas C Geurs, DDS, MS, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham School of Dentistry, Birmingham, Alabama, United States

REFERENCES:
- [Background] Sclar AG. Strategies for management of single-tooth extraction sites in aesthetic implant therapy. J Oral Maxillofac Surg. 2004 Sep;62(9 Suppl 2):90-105. doi: 10.1016/j.joms.2004.06.041. PMID 15332186
- [Background] Lekovic V, Kenney EB, Weinlaender M, Han T, Klokkevold P, Nedic M, Orsini M. A bone regenerative approach to alveolar ridge maintenance following tooth extraction. Report of 10 cases. J Periodontol. 1997 Jun;68(6):563-70. doi: 10.1902/jop.1997.68.6.563. PMID 9203100
- [Background] Lekovic V, Camargo PM, Klokkevold PR, Weinlaender M, Kenney EB, Dimitrijevic B, Nedic M. Preservation of alveolar bone in extraction sockets using bioabsorbable membranes. J Periodontol. 1998 Sep;69(9):1044-9. doi: 10.1902/jop.1998.69.9.1044. PMID 9776033
- [Background] Artzi Z, Tal H, Dayan D. Porous bovine bone mineral in healing of human extraction sockets. Part 1: histomorphometric evaluations at 9 months. J Periodontol. 2000 Jun;71(6):1015-23. doi: 10.1902/jop.2000.71.6.1015. PMID 10914806
- [Background] Artzi Z, Tal H, Dayan D. Porous bovine bone mineral in healing of human extraction sockets: 2. Histochemical observations at 9 months. J Periodontol. 2001 Feb;72(2):152-9. doi: 10.1902/jop.2001.72.2.152. PMID 11288787
- [Background] Froum S, Cho SC, Rosenberg E, Rohrer M, Tarnow D. Histological comparison of healing extraction sockets implanted with bioactive glass or demineralized freeze-dried bone allograft: a pilot study. J Periodontol. 2002 Jan;73(1):94-102. doi: 10.1902/jop.2002.73.1.94. PMID 11846205
- [Background] Zubillaga G, Von Hagen S, Simon BI, Deasy MJ. Changes in alveolar bone height and width following post-extraction ridge augmentation using a fixed bioabsorbable membrane and demineralized freeze-dried bone osteoinductive graft. J Periodontol. 2003 Jul;74(7):965-75. doi: 10.1902/jop.2003.74.7.965. PMID 12931758
- [Background] Iasella JM, Greenwell H, Miller RL, Hill M, Drisko C, Bohra AA, Scheetz JP. Ridge preservation with freeze-dried bone allograft and a collagen membrane compared to extraction alone for implant site development: a clinical and histologic study in humans. J Periodontol. 2003 Jul;74(7):990-9. doi: 10.1902/jop.2003.74.7.990. PMID 12931761
- [Background] Anitua E. Plasma rich in growth factors: preliminary results of use in the preparation of future sites for implants. Int J Oral Maxillofac Implants. 1999 Jul-Aug;14(4):529-35. PMID 10453668
- [Background] Marx RE. Platelet-rich plasma: evidence to support its use. J Oral Maxillofac Surg. 2004 Apr;62(4):489-96. doi: 10.1016/j.joms.2003.12.003. No abstract available. PMID 15085519
- [Background] Nevins M, Giannobile WV, McGuire MK, Kao RT, Mellonig JT, Hinrichs JE, McAllister BS, Murphy KS, McClain PK, Nevins ML, Paquette DW, Han TJ, Reddy MS, Lavin PT, Genco RJ, Lynch SE. Platelet-derived growth factor stimulates bone fill and rate of attachment level gain: results of a large multicenter randomized controlled trial. J Periodontol. 2005 Dec;76(12):2205-15. doi: 10.1902/jop.2005.76.12.2205. PMID 16332231
- [Background] Reddy M, Giannoble E, Nevins M, McGuire M. Kao R, Lynch S. Multicentered radiographic analysis of a regenerative medicine approach to periodontal bone destruction. Southeast Workshop on Tissue Engineering and Biomaterials 2nd Annual February 11-12, 2005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomization was performed by site (teeth) in the mouth. Each participant has only one tooth enrolled in the study.
Units Other Than Participants: teeth
Groups:
- 1 Atraumatic Teeth Extraction: Teeth extraction followed by natural healing
  AtraumaticTeeth Extraction: Teeth extraction alone, allowed to heal for 2 months followed by implant therapy to the sites
Period: Overall Study
Arm/Group | 1 Atraumatic Teeth Extraction | 2- FDBA/TCP | 3 FDBA/TCP+PRP | 4 FDBA/TCP + PDGF
Started | 9; 9 teeth | 11; 11 teeth | 12; 12 teeth | 9; 9 teeth
Completed | 9; 9 teeth | 11; 11 teeth | 12; 12 teeth | 9; 9 teeth
Not Completed | 0; 0 teeth | 0; 0 teeth | 0; 0 teeth | 0; 0 teeth

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Atraumatic Teeth Extraction | 2- FDBA/TCP | 3 FDBA/TCP+PRP | 4 FDBA/TCP + PDGF | Total
Number analyzed (Participants) | 9 | 11 | 12 | 9 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 11 | 6 | 32
  >=65 years | 2 | 3 | 1 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 9 | 6 | 29
  Male | 4 | 2 | 3 | 3 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 1 | 1 | 6
  White | 8 | 7 | 10 | 8 | 33
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Bone-fill in Grafted Post-extraction Sockets Versus Bone-fill in Non-grafted Post-extraction Sockets
Description: New bone formation in grafted extraction sockets to that of sites healed after 8 weeks of post-extraction.
Time Frame: 2 months
Population: Each participant has only one tooth enrolled.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: teeth
Arm/Group | 1 Atraumatic Teeth Extraction | 2- FDBA/TCP | 3 FDBA/TCP+PRP | 4 FDBA/TCP + PDGF
Number analyzed (Participants) | 9 | 11 | 12 | 9
Number analyzed (teeth) | 9 | 11 | 12 | 9
mm | 0.43 (0.24) | 0.27 (0.07) | 0.36 (0.15) | 0.28 (0.09)

ADVERSE EVENTS:
Time Frame: baseline to 2 months
Arm/Group | 1 Atraumatic Teeth Extraction | 2- FDBA/TCP | 3 FDBA/TCP+PRP | 4 FDBA/TCP + PDGF
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11 | 0/12 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11 | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11 | 0/12 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT00641316/Prot_SAP_000.pdf